CLINICAL TRIAL: NCT02225262
Title: Prospective Evaluation of CyberKnife Stereotactic Radiosurgery for Low and Intermediate Risk Prostate Cancer: Emulating Homogenous Dose Distribution
Brief Title: A Phase II Trial of CyberKnife Stereotactic Radiosurgery to Prostate Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Community Cancer Center, Normal, Illinois (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CK Prostate-01
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer; Cancer of the Prostate; Prostate Neoplasm
Keywords: Prostate cancer; CyberKnife; Stereotactic; Radiation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CyberKnife Radiosurgery (Experimental)
  Interventions: Radiation: CyberKnife Radiosurgery

INTERVENTIONS:
Radiation: CyberKnife Radiosurgery — 36.25 Gy delivered in 5 fractions of 7.25 Gy per fraction
  Other Names: CyberKnife

SUMMARY:
The purpose of this study is to determine the effects of CyberKnife radiosurgery in patients with early stage prostate cancer.

The investigators hypothesize that hypofractionated stereotactic radiotherapy via the CyberKnife® can deliver tumor ablating doses of radiation to prostate tumors safely and effectively while sparing the adjacent tissues (rectum, bladder, ureters, urethra, penile bulb, and bowel) from receiving damaging doses of radiation.

DETAILED DESCRIPTION:
The CyberKnife system is a type of radiation machine that uses a special system to precisely focus large doses of x-rays (radiation) on the tumor. The device is designed to concentrate large doses of radiation onto the tumor so that injury from radiation to the nearby normal tissue will be minimal.

ELIGIBILITY:
Inclusion Criteria:

* Male Age ≥ 21
* Histologically proven prostate adenocarcinoma
* Clinical stage T1b-T2b, N0-Nx, M0-Mx (AJCC 6th Edition)
* PSA ≤ 20 ng/ml
* Prostate volume ≤ 100 cc

Patients belonging in one of the following risk groups:

* Low:

  * CS T1b-T2a and Gleason 2-6 and PSA ≤ 10
* Intermediate:

  * CS T2b and Gleason 2-6 and PSA ≤ 10, OR
  * CS T1b-T2b, and Gleason 2-6 and PSA ≤ 20 ng/ml OR Gleason 7 and PSA ≤ 10 ng/ml

Exclusion Criteria:

* Any histology other than adenocarcinoma
* Age < 21
* KPS <= 40 <70
* ECOG Performance Status ≥ 2
* Patient weight >350 lbs. (table limitation)
* Prior XRT to prostate or lower pelvis
* Prior surgery or cryotherapy to prostate
* Implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery, in the investigator's opinion
* Chemotherapy for a malignancy in the last 5 years
* History of an invasive malignancy (other than this prostate cancer, or basal or squamous skin cancers) in the last 5 years
* Hormone ablation for 2 months prior to enrollment, or during treatment

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Local control rate | 5-10 years
  * To assess the effects of hypofractionated stereotactic radiosurgery on the long-term local tumor control of prostate cancer (through documentation of the rate of biochemical Disease-Free Survival [bDFS], Phoenix and ASTRO definitions, at 5 and 10 years).
  * To document the rates of acute and late grade 3-5 gastrointestinal and genitourinary toxicity observed during the years following CyberKnife SRS for prostate cancer.

SECONDARY OUTCOMES:
Overall survival | 5-10 years
  To measure the following in the study population: rates of local failure, distant failure, disease-free survival, disease-specific survival; quality of life (QOL) in generic and organ-specific domains.

CONTACTS AND LOCATIONS:
Overall Officials: Shermian Woodhouse, MD, Principal Investigator — Community Cancer Center
Locations (1):
- Community Cancer Center, Normal, Illinois, United States